CLINICAL TRIAL: NCT01678144
Title: Evaluation of the Safety and Performance of the Medtentia Mitral Valve Repair System When Used in Adults Undergoing Mitral Valve Repair Surgery
Brief Title: Study on Safety and Performance of Medtentia Mitral Valve Repair System in Surgical Repair of Mitral Regurgitation
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Strategic decision by Sponsor
Sponsor: Medtentia International Ltd Oy (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2010-040
Record Dates: First submitted 2012-08-30; First posted 2012-09-03 (Estimated); Results first posted 2019-08-09 (Actual); Last update posted 2019-08-09 (Actual); Status verified 2019-06

CONDITIONS: Mitral Regurgitation; Mitral Insufficiency
Keywords: mitral valve; mitral surgery; mitral repair; mitral annuloplasty; mitral valve surgery; mitral valve repair; mitral valve annuloplasty
MeSH Terms: conditions — Mitral Valve Insufficiency

STUDY DESIGN:
Intervention Model Description: Prospective, multi-national, multi-center, open-label, single-arm
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Medtentia Annuloplasty Ring (MAR) (Experimental): All eligible patients underwent surgical mitral valve repair using annuloplasty device - Medtentia Annuloplasty Ring (MAR)
  Interventions: Device: Mitral valve repair using the Medtentia Annuloplasty Ring (MAR)

INTERVENTIONS:
Device: Mitral valve repair using the Medtentia Annuloplasty Ring (MAR)

SUMMARY:
The purpose of the trial is to demonstrate the safety and performance of the Medtentia Annuloplasty Ring (MAR) during mitral valve repair surgery. In addition, the trial aims to demonstrate that the MAR fulfills the requirements for mitral valve annuloplasty rings.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the safety and performance of the MAR in patients with mitral regurgitation requiring either isolated mitral valve annuloplasty or mitral valve annuloplasty concomitantly with any of the following, either individually or in combination:

* Tricuspid valve repair
* Coronary artery bypass grafting (CABG)
* Valve resection and chordae repair
* Correction of atrial septal defect
* Correction of patent foramen ovale
* Ablation therapy for atrial defibrillation

ELIGIBILITY:
Inclusion criteria:

Eligible patients must meet all the following inclusion criteria:

1. Signed Informed Consent Form.
2. Male or female aged ≥18 to ≤ 85 years on the day of screening. Females of childbearing potential (not surgically sterilized or more than one year post-menopausal) must have a negative pregnancy test (serum beta-human chorionic gonadotropin (beta-hCG) or urine) within 24 hours prior to mitral valve surgery.
3. Patient must meet one of the following indications for mitral repair surgery according to the European Society of Cardiology (ESC) and the American Heart Association (AHA) guidelines, and must have consented to have such surgery before undergoing the informed consent process for this study.

   * Symptomatic patient with chronic severe primary mitral regurgitation (MR), left ventricle ejection fraction (LVEF) > 30% and left ventricle end systolic diameter (LVESD) < 55 mm or
   * Asymptomatic patient with chronic severe primary MR who either:

     * Has LV dysfunction (LVEF ≤ 60 % and/or LVESD ≥ 40 mm or
     * Has a preserved LV function (LVEF> 60% and LVESD < 40 mm) together with a likelihood of a successful and durable repair of > 95 % and an expected mortality rate of < 1% or
     * Has a flail leaflet and LVESD ≥ 40 mm together with a high likelihood of durable repair and a low surgical risk or
     * Has a new onset of atrial fibrillation or pulmonary hypertension (systolic pulmonary pressure > 50 mm Hg at rest) or
   * Asymptomatic patient with chronic moderate or severe primary MR who is to undergo cardiac surgery for another indication when the mitral valve (MV) repair can be performed concomitantly
   * Patient with chronic severe or moderate secondary MR and an LVEF > 30 % who is undergoing CABG concomitantly
4. Patient must have a life expectancy of more than 24 months at the time of screening, assuming they undergo mitral valve annuloplasty.
5. Patient must have a mitral valve diameter corresponding to MAR size 26 - 40 and leaflet thickness (smallest helix height - largest helix height) for which an appropriate MAR ring is available.
6. Patient must be able and willing to attend all scheduled visits and comply with all study procedures.

Exclusion criteria:

Eligible patients must not meet any of the following exclusion criteria:

1. Have had previous cardiac surgery, including but not limited to any of the following: minimally invasive surgery, mitral valve surgery or valvuloplasty, implantation of a prosthetic heart valve or cardiac defibrillator.
2. Have ejection fraction below 30%.
3. Plan to have any concomitant cardiac surgery or procedure other than CABG, tricuspid valve repair, correction of atrial septal defect, closure of auricular appendage, correction of patent foramen ovale and/or ablation therapy for correction of atrial fibrillation performed with the mitral valve repair, which may also include leaflet resection and chordae replacement.
4. Have any structural hindrance or heart abnormality that would make use of the MAR technically infeasible, such as a mitral valve of an unusual size or leaflet thickness for which a suitable MAR is not available, or an obstruction or other abnormality that blocks positioning of the MAR. (Final determination to be made during surgery).
5. Show evidence of having had an acute myocardial infarction (MI) within the 30 days preceding the mitral valve repair surgery.
6. Have a history of stroke within the preceding 12 months or have had any stroke that is not completely clinically resolved and/or significant carotid artery disease (subjects with carotid stenosis ≥50% and/or ulceration).
7. Have recent or evolving bacterial endocarditis or be undergoing antibiotic therapy.
8. Have restricted mobility of the mitral apparatus that results in a valvular area less than 3.0 cm2.
9. Be in need of annular decalcification.
10. Have any comorbidities or conditions that would be a contraindication to open heart surgery or that would place the patient at an unacceptable surgical risk, such as: severe chronic obstructive pulmonary disease (COPD); hepatic failure; immunosuppressive abnormalities or other immunological deficiencies including being immunocompromised or having an autoimmune disease; chronic renal failure requiring dialysis; hematological abnormalities including a history of bleeding diathesis or coagulopathy; being unable to follow the locally recommended anticoagulant regimen; an intolerance or hypersensitivity to anesthetics; cancer that requires further radiation, chemotherapy or surgical treatment.
11. Have a contraindication to trans-esophageal echocardiography (TEE)/ Doppler.
12. Have any recent psychiatric disorder, including drug or alcohol abuse, that in the Investigator's opinion could impair the patient's compliance with study procedures.
13. Be currently or have in the preceding 30 days participated in any other study involving an investigational drug or device.
14. Be an employee of the investigational site directly affiliated with this study, the sponsor or the clinical research organization or have an immediate family member who is.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2011-06-30 (Actual); Primary Completion 2014-07-30 (Actual); Study Completion 2016-04-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kalervo Werkkala, M.D., Prof., Principal Investigator — Helsinki University Central Hospital
Locations (1):
- Helsinki University Hospital, Cardiovascular and Thorax Surgery Clinic, Helsinki, Finland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Konerding MA, Simpanen J, Ihlberg L, Aittomaki J, Werkkala K, Delventhal V, Ackermann M. Comparison of the novel Medtentia double helix mitral annuloplasty system with the Carpentier-Edwards Physio annuloplasty ring: morphological and functional long-term outcome in a mitral valve insufficiency sheep model. J Cardiothorac Surg. 2013 Apr 8;8:70. doi: 10.1186/1749-8090-8-70. PMID 23566678
- [Background] Jensen H, Simpanen J, Smerup M, Bjerre M, Bramsen M, Werkkala K, Vainikka T, Hasenkam JM, Wierup P. Medtentia double helix mitral annuloplasty system evaluated in a porcine experimental model. Innovations (Phila). 2010 Mar;5(2):114-7. doi: 10.1097/IMI.0b013e3181d84316. PMID 22437358
- See also: Medtentia Company Webpage — https://medtentia.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All patients were enrolled at Helsinki University Central Hospital from June 2011 to April 2014.
  During Stage 1 (2011-2012) and Stage 2 (2013-2016) MAR was implanted for 12 patients.
  11 of 24 consented patients did not receive MAR due to non-anatomical fit (majority in Stage 1); for 1 patient MAR was replaced before the operation was completed.
Pre-assignment Details: Patients qualifying for mitral valve repair surgery according to guidelines from the European Society of Cardiology (ESC) and the American Heart Association (AHA) and meeting pre-operative selection criteria.
  Successful implantation rate improved significantly during Stage 2 after sizing adjustment of the implant (Regular and Expanded).
Units Other Than Participants: MAR implant
Period: Stage 1: MAR Classic
Arm/Group | Medtentia Annuloplasty Ring (MAR)
Started | 7; 7 MAR implant
Completed | 6; 6 MAR implant
Not Completed | 1; 1 MAR implant
Not completed — Adverse Event | 1
Period: Stage 2: MAR Regular and MAR Expanded
Arm/Group | Medtentia Annuloplasty Ring (MAR)
Started | 5; 5 MAR implant
Completed | 5; 5 MAR implant
Not Completed | 0; 0 MAR implant

BASELINE CHARACTERISTICS:
Population: Baseline data are provided for patients enrolled in the Stage 1 and Stage 2.
Groups:
- Medtentia Annuloplasty Ring (MAR): Mitral valve repair using the Medtentia Annuloplasty Ring (MAR)
  Mitral valve repair using the Medtentia Annuloplasty Ring (MAR)
Arm/Group | Medtentia Annuloplasty Ring (MAR)
Number analyzed (Participants) | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 5
  >=65 years | 7
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.5 (8.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 9
Region of Enrollment [Number; unit: participants]
  Finland | 12
New York Heart Association (NYHA) Functional Capacity [Number; unit: participants] — Four classes describing the effect of cardiac disease on physical activity: Class I - disease does not limit activity; Class II - slight limitation; Class III - marked limitation; Class IV - inability to carry out any physical activity without discomfort
  participants
    Class I | 2
    Class II | 5
    Class III | 4
    Class IV | 1
Left Ventricular Inner Dimension Systole [Median (Inter-Quartile Range); unit: millimeters] — The dimension of inner edge to inner edge, perpendicular to the long axis of the left ventricle, at the level of the mitral valve leaflet tips, measured at end-systole by trans-thoracic echocardiography. Population: Assessment not available for one patient.
  millimeters
    number analyzed (Participants) | 11
    (all) | 46 [42 to 51]
Mitral valve regurgitation [Number; unit: participants] — Mitral regurgitation according to American College of Cardiology/ American Heart Association (ACC/AHA) classification determined by echocardiography: Class I - trivial (<0.2 cm2 effective regurgitant orifice (ERO)), Class II - mild (0.2-0.29 cm2 ERO), Class III - moderate (0.3-0.39 cm2 ERO), Class IV - severe (≥0.4 cm2 ERO). Population: Assessment not available for one patient.
  participants
    Class I: number analyzed (Participants) | 11
    Class I | 0
    Class II: number analyzed (Participants) | 11
    Class II | 0
    Class III: number analyzed (Participants) | 11
    Class III | 0
    Class IV: number analyzed (Participants) | 11
    Class IV | 11
Smoking status [Count of Participants; unit: Participants]
  Current smoker | 1
  Non-smoker/ Former smoker | 11
Mitral valve leaflet coaptation height [Median (Inter-Quartile Range); unit: millimeters] — Mitral valve leaflet coaptation height assessment by trans-thoracic echocardiography. Population: Assessment not available for one patient.
  millimeters
    number analyzed (Participants) | 11
    (all) | 14 [9.8 to 20]
Left Ventricular Inner Dimension Diastole [Median (Inter-Quartile Range); unit: millimeters] — The dimension of inner edge to inner edge, perpendicular to the long axis of the left ventricle, at the level of the mitral valve leaflet tips, measured at end-diastole by trans-thoracic echocardiography. Population: Assessment not available for one patient.
  millimeters
    number analyzed (Participants) | 11
    (all) | 60 [54 to 63]

OUTCOME MEASURES:

1. Primary Outcome: Safety: All-cause Mortality Occurring in the Time From Surgery Through Hospital Discharge.
Time Frame: Time from surgery through hospital discharge, up to 7 days.
Measure: Count of Participants; unit: Participants
Groups:
- Medtentia Annuloplasty Ring (MAR): Mitral valve repair using the Medtentia Annuloplasty Ring (MAR)
Arm/Group | Medtentia Annuloplasty Ring (MAR)
Number analyzed (Participants) | 12
Participants | 0

2. Primary Outcome: Performance: Percentage of Participants With Improvement by at Least 2 Mitral Regurgitation Classes From Baseline (SC) to Three Months (V03) as Measured by Trans-thoracic Echocardiography (TTE).
Description: Success will be defined as an improvement in at least 2 degrees in mitral regurgitation (MR) class as described in the ACC/AHA Guidelines for the Management of Patients with Valvular Heart Disease (Bonow, et al., 2008).
Time Frame: Time from baseline through V03 (3 months)
Measure: Mean (95% Confidence Interval); unit: percentage of participants
Arm/Group | Medtentia Annuloplasty Ring (MAR)
Number analyzed (Participants) | 11
percentage of participants | 90.91 [58.72 to 99.77]

3. Secondary Outcome: Safety: 30-day Mortality and Mortality at 3 Months, 6 Months, 1 Year, 1.5 Years and 2 Years.
Description: Mortality rates determined both for all-cause mortality and for related deaths only. For the former, the causality status will be determined by the Investigator, and all deaths that are clearly unrelated to the device, the surgery or the underlying medical condition will be excluded from the analysis.
Time Frame: 30 days, 3 months, 6 months, 1 year, 1.5 years and 2 years after surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Medtentia Annuloplasty Ring (MAR)
Number analyzed (Participants) | 12
Participants | 0

4. Secondary Outcome: Safety: The Occurrence, Frequency and Timing of Treatment-emergent Major Adverse Cardiac Events (MACEs).
Description: MACE is defined as stroke and clinically significant myocardial infarction (MI), from surgery to end of study.
Time Frame: From surgery to end of study (2 years)
Measure: Number; unit: Events
Arm/Group | Medtentia Annuloplasty Ring (MAR)
Number analyzed (Participants) | 12
Events | 1

5. Secondary Outcome: Safety: The Occurrence, Nature and Frequency of Treatment-emergent Adverse Events (AEs), in Particular Severe Serious Adverse Device Effects (SADEs).
Description: All the adverse events reported were non-device related.
Time Frame: From surgery to end of study (2 years).
Population: Due to the smaller than planned patient group size the descriptive statistics was used. Adverse events data is presented in Adverse Events section.
Measure: Number; unit: Events
Arm/Group | Medtentia Annuloplasty Ring (MAR)
Number analyzed (Participants) | 12
Events | 30

6. Secondary Outcome: Safety: The Occurrence, Nature and Frequency of Device Deficiencies and Adverse Device Effects (ADEs).
Time Frame: From surgery to end of study (2 years).
Measure: Number; unit: Events
Arm/Group | Medtentia Annuloplasty Ring (MAR)
Number analyzed (Participants) | 12
Events | 0

7. Secondary Outcome: Safety: The Occurrence, Frequency and Nature of Abnormalities in the Period From Surgery Through Follow-up (Detailed List in Description Field).
Description: The occurrence, frequency and nature of abnormalities in any of the following:
  * physical examination
  * vital signs
  * electrocardiography (ECG)
  * echocardiography (ECHO)
  * Laboratory tests
  * Chest X-rays (taken only when clinically indicated)
Time Frame: From surgery to end of study (2 years).
Population: The study was terminated prematurely. Due to the smaller than planned patient group size no sufficient data was collected for planned analysis of this endpoint.
Arm/Group | Medtentia Annuloplasty Ring (MAR)
Number analyzed (Participants) | 0

8. Secondary Outcome: Performance: Mitral Regurgitation (MR) as Seen in Trans-esophageal Echocardiography (TEE) Performed During Surgery Before and After Annuloplasty.
Description: Success will be defined as no or only residual mitral regurgitation (MR).
Time Frame: Day of surgery visit (V01).
Population: The data for this outcome measure was not collected.This was a part of the echocardiography investigation protocol and therefore was not documented on electronic case report form although the surgeon in charge performed the investigation on the operation table.
Arm/Group | Medtentia Annuloplasty Ring (MAR)
Number analyzed (Participants) | 0

9. Secondary Outcome: Performance: Percentage of Participants With Improvement by at Least 2 Mitral Regurgitation Classes at Each Follow-up Visit (V04-V06) of the Improvement in MR From Screening, as Measured by Trans-thoracic Echocardiography (TTE).
Description: Measurement analysis at 24 months after successful MAR implantation.
Time Frame: V06 (24 months)
Population: The study was terminated prematurely. Due to the smaller than planned patient group size no patient data at V04 (6 months) and V05 (12 months) was analyzed for this endpoint. The results provided are only for V06 (24 months).
Measure: Mean (95% Confidence Interval); unit: percentage of participants
Arm/Group | Medtentia Annuloplasty Ring (MAR)
Number analyzed (Participants) | 11
percentage of participants | 100 [71.51 to 100]

10. Other Pre Specified Outcome: Exploratory: Change in the Mitral Regurgitation (MR) Parameters, as Measured Using TTE.
Description: Change from screening at each follow-up visit in the following MR parameters, as measured using TTE:
  * Left ventricular inner dimension systole and diastole assessment by trans-thoracic echocardiography (the dimension of inner edge to inner edge, perpendicular to the long axis of the left ventricle, at the level of the mitral valve leaflet tips, measured at end-systole and end-diastole)
  * Coaptation height
Time Frame: From screening to end of study (up to 2 years)
Population: The outcome is reported for subjects and follow up visits where data is available
Measure: Median (Inter-Quartile Range); unit: millimeters
Arm/Group | Medtentia Annuloplasty Ring (MAR)
Number analyzed (Participants) | 11
millimeters
  Left Ventricular Inner Dimension Systole 3 months | 40 [34 to 43]
  Left Ventricular Inner Dimension Systole 2 years | 38 [36 to 43]
  Left Ventricular Inner Dimension Diastole 3 months | 50 [45 to 56]
  Left Ventricular Inner Dimension Diastole 2 years | 51 [49 to 52]
  Coaptation Height 3 months: number analyzed (Participants) | 10
  Coaptation Height 3 months | 6.2 [2.7 to 12.7]
  Coaptation Height 2 years: number analyzed (Participants) | 9
  Coaptation Height 2 years | 7.3 [3.6 to 11]

11. Other Pre Specified Outcome: Exploratory: Duration of the Key Stages of the Annuloplasty Procedure.
Description: Duration of the following key stages of the annuloplasty procedure:
  * MAR implantation time (beginning with the measurement of the annulus size and ending with the completion of the last suture, but not including the time needed to measure leaflet thickness)
  * MAR rotation time
  * Suturing time (from start of annulus suturing until last knot)
  * Aortic clamp time
  * Cardiac arrest time
Time Frame: Day of surgery visit (V01)
Population: MAR rotation time assessment available for 9 patients only.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Medtentia Annuloplasty Ring (MAR)
Number analyzed (Participants) | 11
minutes
  Aortic clamp time | 87.2 (24.5)
  MAR implantation time | 16.9 (5.0)
  Suturing time | 14.6 (4.1)
  MAR rotation time: number analyzed (Participants) | 9
  MAR rotation time | 2.5 (1.4)
  Cardiac arrest time | 116.2 (32.8)

12. Other Pre Specified Outcome: Exploratory: Changes From Screening in NYHA Classification at All Follow-up Visits Except Discharge.
Time Frame: At screening and at each follow-up visit (except for discharge visit, up to 2 years).
Measure: Count of Participants; unit: Participants
Arm/Group | Medtentia Annuloplasty Ring (MAR)
Number analyzed (Participants) | 11
Participants
  3 monts: Class I | 8
  3 monts: Class II | 3
  3 monts: Class III | 0
  3 monts: Class IV | 0
  6 months: Class I | 9
  6 months: Class II | 2
  6 months: Class III | 0
  6 months: Class IV | 0
  1 year: Class I | 10
  1 year: Class II | 1
  1 year: Class III | 0
  1 year: Class IV | 0
  2 years: Class I | 11
  2 years: Class II | 0
  2 years: Class III | 0
  2 years: Class IV | 0

13. Other Pre Specified Outcome: Exploratory: Thickness of the Anterior Leaflet Segment A2 and the Posterior Scallop P2 of the Mitral Valve (MV) Leaflets, as Measured With the Dedicated Medtentia Leaflet Measurement Tool.
Time Frame: Day of surgery visit (V01)
Population: The leaflet measuring tool was designed to compress the leaflet between two jaws to measure the thickness. Due to soft tissue getting compressed between these two jaws the measure was not seen accurate, therefore this procedure was omitted in the study.
Arm/Group | Medtentia Annuloplasty Ring (MAR)
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: AEs documented from the point of surgery trough the follow-up (2 years).
Description: Common episodes during surgery (e.g. blood loss) and postoperative (e.g. pain, nausea, normal bruising) that are not considered clinically relevant by the Investigator should not be captured as AEs unless the event is worse than would normally be expected.
  Cases of excessive or abnormal bleeding or blood loss should be reported as AEs. Normal surgery-related laboratory test fluctuations common after surgery and not usually considered clinically significant are not considered to be AEs.
Arm/Group | Medtentia Annuloplasty Ring (MAR)
All-Cause Mortality (participants affected / at risk) | 0/12
Serious Adverse Events (participants affected / at risk) | 7/12
Other Adverse Events (participants affected / at risk) | 8/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Medtentia Annuloplasty Ring (MAR) (N=12)
Residual mitral regurgitation leading to re-operation (Cardiac disorders) | 1 (1)
Takotsubo cardiomyopathy (Cardiac disorders) | 1 (1)
Peritonsilitis l.dx (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Postoperative delirium (Psychiatric disorders) | 1 (1)
Atrial fibrillation worsening (Cardiac disorders) | 1 (1)
Postoperative fever (Injury, poisoning and procedural complications) | 1 (1)
Increased white blood cell count (Investigations) | 1 (1)
Transient ischemic attack (Nervous system disorders) | 1 (1)
Urinary tract infection/ urosepsis (Infections and infestations) | 1 (1)
Pre-symptomatic migraine (Nervous system disorders) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 2 (2)
Atrial flutter (Cardiac disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Medtentia Annuloplasty Ring (MAR) (N=12)
Atrial fibrillation worsening (Cardiac disorders) | 2 (2)
Atrial fibrillation (Cardiac disorders) | 4 (5)
Atrial flutter (Cardiac disorders) | 2 (2)
Urinary tract infection (Infections and infestations) | 1 (1)
Wound infection (Infections and infestations) | 2 (2) — Reported adverse event terms: Wound infection, left leg donor site and Minor wound infection.
Asthma bronchiale (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Ventricular tachycardia episode (Cardiac disorders) | 1 (1)
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Common cold (Infections and infestations) | 1 (1)

LIMITATIONS AND CAVEATS:
The study was terminated prematurely. The smaller than planned patient group size did not allow testing the study hypothesis in full. Due to the limited number of patients only descriptive statistics were used.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less